CLINICAL TRIAL: NCT06561919
Title: STIMPulseControl Ancillary Speech Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Steffen Paschen (Other)
Collaborators: Czech Technical University in Prague (Other); Insel Gruppe AG, University Hospital Bern (Other); Philipps University Marburg (Other); University Hospital Schleswig-Holstein (Other); Amsterdam University Medical Centers (UMC), Location Academic Medical Center (AMC) (Other)
Responsible Party: Sponsor-Investigator, Steffen Paschen, MD, University of Kiel
Organization: University of Kiel (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KKS-313-A
Record Dates: First submitted 2024-06-24; First posted 2024-08-20 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease; Impulse Control Disorder
Keywords: Speech
MeSH Terms: conditions — Parkinson Disease; Disruptive, Impulse Control, and Conduct Disorders; Speech

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DBS-group (Other): Within indication and clinical routine: bilateral high frequency deep brain stimulation of the subthalamic necleus combined with best medical treatment
  Interventions: Procedure: bilateral high frequency deep brain stimulation of the subthalamic neucleus combined with best medical treatment according to widely accepted expert consensus paper
- BMT-group (Other): Within indication and clinical routine: best medical treatment
  Interventions: Drug: best medical treatment for management of impulse control in Parkinson´s disease according to widely accepted expert consensus paper

INTERVENTIONS:
Procedure: bilateral high frequency deep brain stimulation of the subthalamic neucleus combined with best medical treatment according to widely accepted expert consensus paper — Best medical treatment according to widely accepted expert consensus Paper
  Other Names: best medical treatment for manangement of impulse control in Parkinson´s disease
  Arms: DBS-group
Drug: best medical treatment for management of impulse control in Parkinson´s disease according to widely accepted expert consensus paper — Best medical treatment according to widely accepted consensus Paper
  Arms: BMT-group

SUMMARY:
Speech assessment is a substudy to the STIMPulseControl study (hereinafter referred to as the main study), where audio recordings of patients voices will be recorded as part of a speech analysis in the main study, for this optional ancillary study.

DETAILED DESCRIPTION:
Speech of all study patients enrolled in the STIMPulseControl main study will be recorded at three points of time in a standardized way. Following this ancillary protocol, patients speech will be recorded at the baseline visit (preoperatively), at the 6-months visit and at the 12-months visit postoperatively.

For the baseline speech assessment the same protocol will be performed in chronic medication conditions. At 12-month follow up, we will repeat the speech protocol in chronic medication and stimulation condition. The recordings will be done in each centre in a decentralized way and the audio files will be produced according to a standardized protocol, and assisted by a step-by-step guided speech recording software.

Main aims and hypothesis for automated speech analysis study are safety measures for surgical interventions in PD assessment of parkinsonian (hypokinetic) motor speech features outcome after STN-DBS, assessment of dyskinetic (hyperkinetic) motor speech features outcome after STN-DBS, assessment of capsular speech features outcome after STN-DBS in PD emotional and cognitive speech outcomes to be used in surgical and pharmacological interventions in PD assessment of acoustic and linguistic speech features as proxy for behaviour and cognitive changes in PD, comparison of emotional and cognitive speech outcomes before and 1-year after STN-DBS + BMT vs BMT alone.

ELIGIBILITY:
Inclusion Criteria:

Please refer to main study (STIMPulseControl KKS-313)

Exclusion Criteria:

Please refer to main study (STIMPulseControl KKS-313)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2027-07-15 (Estimated); Study Completion 2028-07-15 (Estimated)

PRIMARY OUTCOMES:
Titel: PART 1: Assessment of parkinsonian motor speech features (hypokinetic dysarthria) outcome after STN-DBS | 12 months
  primary aim: To globally assess motor speech features of PD change after STN-DBS intervention.
  Outcome: A compound score resulting from the normalized average of the main speech domains of hypokinetic dysarthria (i.e.phonation, articulation, prosody and timing) will be analyzed.
  For example, as proxy of phonation/voice quality, harmonics-to-noise ratio will be used. For the assessment of articulation changes, voice to onset (VOT) and Resonant frequency attenuation (RFA) will be assessed. Monopitch, will be assessed using the standard deviation of fundamental frequency (sdF0), while reduced intensity of speech variability or monoloudness will be assessed using the standard deviation of speech intensity (sdInt). To assess timing abnormalities seen in PD, prolonged pauses (PrLP), disrupting natural rhythm of speech, will be used.
Titel PART 2: Assessment of acoustic and linguistic speech features as proxy for behavior and cognitive changes in PD | 12 months
  primary aim: To assess how paralinguistic speech content changes after STN-DBS intervention.
  Outcome: A compound score resulting from the normalized average of the main emotional paralinguistic features (such as pitch variability; duration of voiced segments, pause durations and intensity variability).
Titel PART 2: Assessment of acoustic and linguistic speech features as proxy for behavior and cognitive changes in PD | 12 months
  primary aim: To assess how semantic speech content changes after STN-DBS intervention.
  Outcome: A compound score resulting from the normalized average of the main semantic features (such as content density, N-grams parameter, or moving-average type-token ratio).

SECONDARY OUTCOMES:
PART I/B: Safety measures for surgical interventions in PD | 12 months
  secondary aim B: Comparison of paralinguistic speech outcomes before and 1-year after STN-DBS + BMT vs BMT alone.
  Outcome: Comparison of the rate of change of the compound score resulting from the normalized average of the main semantic features (such as content density, N-grams parameter, or moving-average type-token ratio).
PART I/B: Safety measures for surgical interventions in PD | 12 months
  secondary aim B: Comparison of semantic speech outcomes before and 1-year after STN-DBS + BMT vs BMT alone.
  Outcome: Comparison of the rate of change of the compound score resulting from the normalized average of the main semantic features (such as content density, N-grams parameter, or moving-average type-token ratio).
PART II/C: Emotional and cognitive speech outcomes to be used in surgical and pharmacological interventions in PD | 12 months
  secondary aim C: Assessment of capsular speech features outcome after STN-DBS in PD.
  Outcome: A compound score resulting from the normalized average of the main speech features affected by capsular stimulation induced side-effects (such as net speech rate and pitch breaks during sustained phonation).
PART I/A: Safety measures for surgical interventions in PD | 12 months
  secondary aim A: Assessment of dyskinetic (hyperkinetic) motor speech features outcome after STN-DBS.
  Outcome: A compound score resulting from the normalized average of the main speech features affected by dyskinesia (such as intensity variability, breading capacity and spectral features variability).

CONTACTS AND LOCATIONS:
Overall Officials: Jan Rusz, Prof., Study Chair — Czech Technical Iniversity in Prague, Faculty of Electrical Engineering
Locations (12):
- Germany (9):
  - University Hospital Cologne, Cologne
  - University Hospital Carl Gustav Carus, Dresden
  - University Hospital Duesseldorf, Düsseldorf
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - University Hospital Schleswig-Holstein (UKSH), Campus Kiel, Kiel
  - University Hospital of Giessen and Marburg (UKGM), Campus Marburg, Marburg
  - Charité Campus Mitte, Mitte
  - University Hospital Tuebingen, Tübingen
  - University Hospital Wuerzburg, Würzburg
- Amsterdam University Medical Center, Amsterdam, Netherlands
- Switzerland (2):
  - University Hospital of Bern (Inselspital), Bern
  - University Hospital Zuerich (USZ), Zurich

IPD SHARING:
Plan to Share IPD: No